CLINICAL TRIAL: NCT03374319
Title: Somatotopic Configuration of Distal Residual Limb Tissues in Lower Extremity Amputations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Matthew Carty, Staff Surgeon, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014p001379; CDMRP-160165 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2017-09-18; First posted 2017-12-15 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Modified amputation procedure
  Interventions: Procedure: Modified amputation procedure

INTERVENTIONS:
Procedure: Modified amputation procedure — A stair-step (BKA) or fishmouth (AKA) incision will be made. Tibial and fibular or femoral osteotomies will be performed. Segments of the tibialis anterior (TA), peroneus longus (PL), lateral gastrocnemius (LG) and tibialis posterior (TP) muscles will be isolated, as well as the quadriceps (Q) and hamstring (H) groups in the AKA model; if it is not possible to preserve native innervation to these muscles, functional motor units will be constructed from muscle coapted to the appropriate motor nerve endings. The distal tibial and peroneal nerves will be redirected to skin patches in the distal or proximal thigh. Coaptation of the TA/LG, PL/TP and Q/H muscles will then be performed to promote dynamic coupling of these agonist/antagonist pairs. The skin envelope will then be closed in layers over percutaneous drains.
  Other Names: Ewing; AMI; agonist-antagonist myoneural interface

SUMMARY:
The hypothesis of this research protocol is that we will be able to redesign the manner in which lower limb amputations are performed so as to include biological actuators that will enable the successful employment of next generation lower extremity prostheses. The specific aims of the project are as follows:

1. To define a standardized approach to the performance of a novel operative procedure for both below knee (BKA) and above knee (AKA) amputations
2. To measure the degree of volitional motor activation and excursion achievable in the residual limb constructs, and to determine the optimal configuration and design of such constructs
3. To describe the extent of proprioceptive and other sensory feedback achievable through the employment of these modified surgical techniques
4. To validate the functional and somatosensory superiority of the proposed amputation technique over standard approaches to BKA and AKA
5. To develop a modified acute postoperative rehabilitation strategy suited to this new surgical approach

DETAILED DESCRIPTION:
Historical Background

Lower extremity amputation is among the oldest known surgical procedures in medical history. Despite the passage of over two millennia, however, relatively little has changed in the operative approach. Currently, lower limb amputation is indicated most frequently for lower extremity compromise due to severe peripheral vascular disease, followed in short order by trauma, tumors, infections and congenital limb deficiencies. Estimates of frequency of lower limb amputations range from 30,000-40,000 cases per year in the United States alone.

Normal function of the lower limb is enabled through the interplay of multiple muscle groups acting in concert. Ambulation is a remarkably orchestrated biomechanical process that is dependent upon a complex feedback loop involving the central and peripheral nervous systems and the musculoskeletal system. In their native state, the muscles of the lower extremity exist in a balanced agonist/antagonist milieu in which volitional activation of one muscle leads not only to its contracture, but also passive stretch of its opposite. Changes in muscle tension manifest through these changes lead to stimulation of specialized receptors within the muscle fibers that transmit joint position information to the cerebral cortex. Such feedback, in conjunction with cutaneous sensory information from skin mechanoreceptors, provides us with a sense of limb proprioception that ultimately enables high fidelity limb control, even in the absence of visual feedback.

However, the standard operative approach to lower limb amputation at either the below knee (BKA) or above knee (AKA) level obliterates many of the dynamic relationships characteristic of the uninjured lower extremity. Initial exposure is accomplished through either a stair-step (BKA) or fishmouth (AKA) pattern incision, followed by progressive transection of muscles, vessels, nerves and bone at the level of the incision. Tissues distal to the site of structural transection are discarded, regardless of whether or not there may be viable segments, and the proximal residual muscles are layered over the distal transected bone in order to provide insulation to this exposed osseous surface. The surrounding skin is then advanced over the bone/muscle infrastructure in order to achieve definitive closure. The rudimentary approximation of tissues in the distal limb in these approaches results in a disorganized scar mass in which normal dynamic muscle relationships are destroyed. The uncoupling of native agonist/antagonist muscle pairings results in isometric contraction of residual muscle groups upon volitional activation, producing incomplete, unbalanced neural feedback to the brain that results in aberrant perception of residual limb position. Such disturbed feedback not only results in impaired ambulatory function with prosthetics, but also manifests as pathological sensory perception of the extremity in the form of phantom limb and phantom pain symptomatology.

To date, providers and patients have tolerated the limitations of these approaches due to the fairly simplistic goal of lower limb amputation: to provide a stable, padded surface for prosthesis mounting. Historically, lower limb prostheses have afforded amputees the opportunity to recover at least some measure of ambulatory function. Standard lower limb prostheses currently afford the wearer the walk in a rudimentary fashion, as well as occasionally run. However, such devices have generally not been able to recapitulate the complex biomechanics of the human lower limb due to limited ranges of motion and lack of feedback control. These limitations have resulted in substantially altered kinematics in lower limb amputees that are associated with derangements in energy expenditure profiles that worsen with laterality and ascending level.

An age is dawning, however, in which the capabilities of modern prostheses are broadening remarkably. Technological advances including increasingly miniaturized electronics, wireless communications and ever-refined positional sensors have enabled prosthetic developers to create next-generation bionic limbs with markedly enhanced degrees of freedom over prior models. Such prostheses have been demonstrated to markedly improve the energy expenditure of amputees who utilize them appropriately. Even more advanced prostheses are currently under development that incorporate the ability to provide active intrinsic limb control to facilitate complex motor actions such as dancing and balancing on one leg. In addition, prototype prosthetics are currently being developed that have the potential to offer sensory feedback - both tactile and positional - in a manner never before witnessed. Such prosthetics, while not yet available commercially, are presently being utilized in experimental settings.

However, these technological advancements in the sphere of prosthesis development have not been matched with surgical advancements with regards to management of the residual limb. Classic techniques to lower limb amputation do not provide innervated interfaces that can serve as relays for complex prosthesis control; without such biological actuators in the residual limb to provide conduits for information exchange, next generation prostheses are of little use. Stated another way, next generation prosthetics currently incorporate drivers and sensors capable of providing far more enhanced functionality than ever before witnessed, but standard approaches to limb amputation do not provide a way of effectively linking these prosthetics to their intended beneficiaries. An evolution in the manner in which lower limb amputations are performed is now required - one that will provide a biological interface that will allow lower limb amputees to take advantage of the enhanced capabilities offered by the remarkable prostheses currently under development.

Previous Pre-Clinical or Clinical Studies

Recognition of the increased need for effective neural interfaces for prosthetic limbs has been evidenced by an expanding number of efforts in this sphere over the past decade. Initial efforts to provide high resolution control of distal prostheses were focused primarily on direct and indirect brain interfaces, either through placement of electroencephalographic scalp sensors or implantable parenchymal electrodes, respectively. However, such endeavors have been plagued by poor resolution, inconsistencies in signal acquisition and progressive foreign body reactions leading to impulse degradation over time.

As the limitations of brain interfaces have become more evident, focus has shifted to direct peripheral nerve interfaces including interposed sieves and cuffs designed to transduce electrical signals directly from individual nerve fascicles to distal prostheses. Such monitors have, however, shown little clinical promise due to progressive nerve compression secondary to scarring, as well as significant neurological crosstalk and interference in biological models.

As such, the most promising efforts regarding peripheral nerve interface development are now within the realm of biological systems. The two leading models in this sphere are as follows:

* Targeted Muscle Reinnervation (TMR): TMR is a technique whereby a series of nerve transfers is utilized to reinnervate specific target muscles to create additional prosthetic control sites after proximal limb amputation. These nerve transfers offer intuitive control of distal prostheses because the reinnervated muscles are controlled by the same nerves that once innervated the amputated limb. Signals created by the residual nerves are amplified by the recipient muscles, which are captured by surface electrodes and transduced to the distal prosthesis. TMR procedures have been performed on more than 40 patients to date. Limitations of this technique, however, include the finite number of available electromyographic signal sites due to anatomic constraints and issues with long-term signal fidelity.
* Regenerative Peripheral Nerve Interfaces (RPNI): RPNI offers an alternative version of an innervated biological interface. An RPNI is a surgical construct that consists of a non-vascularized segment of muscle that is coapted to a distal motor or sensory nerve ending. Unlike TMR, the RPNI muscle is not recruited from an otherwise normally innervated proximal muscle; instead, it is constructed as a free graft from orthotopically sourced donor tissue. The muscle segment is gradually reinnervated by the redirected nerve ending, which then promotes volitional activation of the muscle segment when triggered by the central nervous system. As in TMR, intuitive control occurs because the reinnervated muscles are controlled by the same nerves that once innervated the amputated limb. Unlike TMR, however, there are no limitations on anatomic sites and there does not appear to be problems with long-term signal fidelity.

While both TMR and RPNIs have demonstrated promise in offering improved functionality to patients who have already undergone amputation, neither technique has been incorporated into a fundamental redesign of the way in which amputations are performed in the first place; in all cases of clinical implementation of TMR or RPNIs reported to date in the literature, these techniques have been employed to further optimize the functionality of patients who have already experienced limb loss.

Rationale and Potential Benefits

This clinical protocol proposes an iteration of the RPNI model, with the intent of incorporating these surgical constructs into the design of lower limb amputations at the time of limb sacrifice. Given the success of this technique to date, the investigators believe that incorporation of innervated muscle segments into residual limb design has the potential to provide lower limb amputees with a biological interface for unprecedented prosthetic motor control that is not only high resolution but also highly intuitive and capable of restoring limb proprioception. In addition, it is anticipated that allowing amputees to have greater control of advanced prostheses may offer the potential to normalize gait kinematics, thereby correcting alterations in energy expenditure that have been previously reported. Such measures hold the promise of optimizing the functional and overall health of lower limb amputees, thereby reducing the morbidity currently associated with the amputee status.

Specific Aims

The hypothesis of this research protocol is that we will be able to redesign the manner in which lower limb amputations are performed so as to include biological actuators that will enable the successful employment of next generation lower extremity prostheses. The specific aims of the project are as follows:

1. To define a standardized approach to the performance of a novel operative procedure for both below knee (BKA) and above knee (AKA) amputations
2. To measure the degree of volitional motor activation and excursion achievable in the residual limb constructs, and to determine the optimal configuration and design of such constructs
3. To describe the extent of proprioceptive and other sensory feedback achievable through the employment of these modified surgical techniques
4. To validate the functional and somatosensory superiority of the proposed amputation technique over standard approaches to BKA and AKA
5. To develop a modified acute postoperative rehabilitation strategy suited to this new surgical approach

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 65
* Candidates for elective unilateral or bilateral lower extremity amputation at either the above knee or below knee level due to traumatic injury, congenital limb deformities or progressive arthritis
* Must demonstrate sufficiently sound health to undergo the operative procedure, including adequate cardiopulmonary stability to undergo general anesthesia (specifically, American Society of Anesthesiology Class I or II)
* Must have intact inherent wound healing capacity
* Must demonstrate adequate communication skills to convey the status of their sensorimotor recovery throughout the postoperative phase,
* Must exhibit proper level of motivation to comply with postoperative follow up requirements.

Exclusion Criteria:

* Patients beyond the stated age restrictions
* Those with severe illness rendering them unable to undergo the operative procedure safely (e.g., unresolved sepsis or cardiopulmonary instability manifest as documented coronary artery disease and/or chronic obstructive pulmonary disease).
* Patients with impairment in inherent wound healing pathways, such as those with primary connective tissue disorders or those on chronic steroid therapy
* Patients with extensive peripheral neuropathies (diabetic or otherwise) that would potentially inhibit appropriate reinnervation of the surgical constructs
* Active smokers; those patients willing to undergo tobacco cessation will need to be completely abstinent from tobacco use for at least 6 weeks preoperatively
* Patients who are unable to provide informed consent and those with a demonstrated history of poor compliance
* Pregnant women will not be considered due to the potential risks of general anesthesia.

Patients will not be excluded from participation in the study on the grounds of minority status, religious status, race or gender. Non-English speaking patients will not be excluded from the study; interpreters will be made available to them for translation of both verbal interactions and written documents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Motor Unit Innervation | 0-48 months
  Intact volitional activation of motor constructs, as assessed by electromyographic evidence of activation (muscle potentials measured in mV)
Motor Unit Excursion | 0-48 months
  Intact volitional activation of motor constructs with measurable excursion, as assessed by ultrasound (excursion measured in mm)
Proprioception Recovery | 0-48 months
  Manifestation of functional proprioception with motor unit activation, as evidenced by spatial limb position testing using a modified lower limb prosthesis (accurate limb positioning relative to target measured in mm)

SECONDARY OUTCOMES:
Infection Rate | 0-48 months
  Postoperative infection rate
Delayed Wound Healing Rate | 0-48 months
  Postoperative delayed wound healing rate
Operative Revision Rate | 0-48 months
  Subsequent rate of reoperation
Seroma Rate | 0-48 months
  Postoperative seroma rate
Deep Vein Thrombosis Rate | 0-48 months
  Postoperative deep vein thrombosis rate
30-Day Mortality Rate | 0-48 months
  Postoperative 30-day mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Carty, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Massachusetts Institute of Technology Media Lab, Cambridge, Massachusetts

IPD SHARING:
Plan to Share IPD: No
No plan for individual participant data sharing

REFERENCES:
- [Background] Ziegler-Graham K, MacKenzie EJ, Ephraim PL, Travison TG, Brookmeyer R. Estimating the prevalence of limb loss in the United States: 2005 to 2050. Arch Phys Med Rehabil. 2008 Mar;89(3):422-9. doi: 10.1016/j.apmr.2007.11.005. PMID 18295618
- [Background] Waters RL, Perry J, Antonelli D, Hislop H. Energy cost of walking of amputees: the influence of level of amputation. J Bone Joint Surg Am. 1976 Jan;58(1):42-6. PMID 1249111
- [Background] Herr HM, Grabowski AM. Bionic ankle-foot prosthesis normalizes walking gait for persons with leg amputation. Proc Biol Sci. 2012 Feb 7;279(1728):457-64. doi: 10.1098/rspb.2011.1194. Epub 2011 Jul 13. PMID 21752817
- [Background] Schultz AE, Kuiken TA. Neural interfaces for control of upper limb prostheses: the state of the art and future possibilities. PM R. 2011 Jan;3(1):55-67. doi: 10.1016/j.pmrj.2010.06.016. PMID 21257135
- [Background] Shih JJ, Krusienski DJ, Wolpaw JR. Brain-computer interfaces in medicine. Mayo Clin Proc. 2012 Mar;87(3):268-79. doi: 10.1016/j.mayocp.2011.12.008. Epub 2012 Feb 10. PMID 22325364
- [Background] Kung TA, Bueno RA, Alkhalefah GK, Langhals NB, Urbanchek MG, Cederna PS. Innovations in prosthetic interfaces for the upper extremity. Plast Reconstr Surg. 2013 Dec;132(6):1515-1523. doi: 10.1097/PRS.0b013e3182a97e5f. PMID 24281580
- [Background] Navarro X, Krueger TB, Lago N, Micera S, Stieglitz T, Dario P. A critical review of interfaces with the peripheral nervous system for the control of neuroprostheses and hybrid bionic systems. J Peripher Nerv Syst. 2005 Sep;10(3):229-58. doi: 10.1111/j.1085-9489.2005.10303.x. PMID 16221284
- [Background] Dumanian GA, Ko JH, O'Shaughnessy KD, Kim PS, Wilson CJ, Kuiken TA. Targeted reinnervation for transhumeral amputees: current surgical technique and update on results. Plast Reconstr Surg. 2009 Sep;124(3):863-869. doi: 10.1097/PRS.0b013e3181b038c9. PMID 19730305
- [Background] Kuiken TA, Li G, Lock BA, Lipschutz RD, Miller LA, Stubblefield KA, Englehart KB. Targeted muscle reinnervation for real-time myoelectric control of multifunction artificial arms. JAMA. 2009 Feb 11;301(6):619-28. doi: 10.1001/jama.2009.116. PMID 19211469
- [Background] Li YG, Chen XJ, Zhang YZ, Han DZ, Yan DX, Gao GZ, Zhao XC, Sun WJ. Three-dimensional digitalized virtual planning for retrograde sural neurovascular island flaps: a comparative study. Burns. 2014 Aug;40(5):974-80. doi: 10.1016/j.burns.2013.10.009. Epub 2013 Nov 26. PMID 24290858
- [Derived] Srinivasan SS, Gutierrez-Arango S, Teng AC, Israel E, Song H, Bailey ZK, Carty MJ, Freed LE, Herr HM. Neural interfacing architecture enables enhanced motor control and residual limb functionality postamputation. Proc Natl Acad Sci U S A. 2021 Mar 2;118(9):e2019555118. doi: 10.1073/pnas.2019555118. PMID 33593940